CLINICAL TRIAL: NCT03985631
Title: Tai Chi Intervention by Telerehabilitation as an Innovative Solution for Parkinson's Disease Population
Brief Title: Tai Chi Intervention by Telerehabilitation
Acronym: TeleParkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-3253
Record Dates: First submitted 2019-05-23; First posted 2019-06-14 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: Tai Chi; Telerehabilitation; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Single group receiving the intevention, one evaluation before and 1 one after the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): Tai Chi intervention by telerehabilitation (3-month intervention, three sessions per week: two supervised session and one unsupervised session).
  Interventions: Other: Rehabilitation intervention

INTERVENTIONS:
Other: Rehabilitation intervention — Rehabilitation sessions based on Tai Chi through telerehabilitation
  Other Names: Télérehabilitation (Tai Chi)

SUMMARY:
Rational : A lot of people in the province of Quebec suffer from Parkinson's disease and they are mostly vulnerable because they gradually lose their autonomy with the worsening of the disease. Physiotherapy was proven to be an effective treatment method for these patients. However, accessibility to care remains a major issue.

Objective: This project aims to establish the clinical feasibility of a Tai chi rehabilitation program through tele rehabilitation to patients suffering of Parkinson's disease.

Methodology : This pilot study will be conduct with a pre/post-test device. Therefore, to reach the objective, an evaluation will be done before the intervention and directly after the end of the 12 weeks program. Also, the obstacles encountered during the interventions will be noted in a logbook.

Benefits: This is a priority research because its aim is to develop a care system that is efficient and accessible for a target population. The results of this study will confirm the possibility to put in place a telerehabilitation program who could reach, on a larger scale, more patients suffering from Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with Parkinson Disease according to the " Movement Disorders Society's diagnostic criteria " for at least 3 years
* Presence of a postural instability measured by the pull test according to Movement Disorders Society-Sponsored revision scale of Unified Parkinson Disease Rating scale " (MDS-UPDRS) with a score to item 3, 12 ≥ 1,
* Have access to Internet
* Have a caregiver available during rehabilitation sessions

Exclusion Criteria:

* Have a une cognitive impairment measured by the " Mini-Mental State Examination " (MMSE), with a total score < 24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Change in balance | 3 months
  Mini BESTest

SECONDARY OUTCOMES:
Change in quality of life | 3 months
  PDQ-39 (Parkinson Disease Questionnaire - 39)This questionnaire assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living.Percentage score ranging between 0 and 100 (100%: more health problems).
Satisfaction with service received | 3 months
  Satisfaction with health care services received (questionnaire, total score on 100%, 0% not satisfied at all with service received, 100%: very satisfied) )

CONTACTS AND LOCATIONS:
Overall Officials: Michel Tousignant, PhD, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Université de Sherbrooke, Sherbrooke, Quebec
  - Research Centre on Aging, Sherbrooke

IPD SHARING:
Plan to Share IPD: No